CLINICAL TRIAL: NCT04858152
Title: Autologous Transplantation of Hair Follicles for the Treatment of Vitiligo on Glabrous Skin
Brief Title: Hair Transplantation for Treatment of Vitiligo
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistic issues
Sponsor: Mehdi Rashighi (Other)
Responsible Party: Sponsor-Investigator, Mehdi Rashighi, Principal Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00022455
Record Dates: First submitted 2021-04-09; First posted 2021-04-26 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental Arm: Transplantation of hair follicles to non-hair bearing areas affected by vitiligo (Experimental): Punch biopsies will be used to extract hair follicles from area on participant's body that is not affected by vitiligo and has hair growth. The follicles will then be transplanted into an area of the body affected by vitiligo that is hairless.
  Interventions: Procedure: Follicular Unit Extraction via punch biopsy

INTERVENTIONS:
Procedure: Follicular Unit Extraction via punch biopsy — Follicular unit extraction will be performed using standard 0.7mm - 1mm punch biopsies. The donor site, which will be selected as a vitiligo-free, hair-bearing area that is not visible per patient's preference, will be harvested via punch biopsies and transplanted to the recipient site, which will be the glabrous skin of the hands or feet.

SUMMARY:
There are several surgical methods to treat vitiligo patches, and follicular unit extraction (FUE) is one among them. FUE, performed using punch biopsy extraction and hair follicle transplantation, has proven safe and effective in multiple studies for treatment of hair bearing (non-glabrous) skin. This technique has not yet been trialed on hairless areas (glabrous skin) affected by vitiligo, such as the lips, fingertips, knuckles, wrists, and feet, which tend to be resistant to standard treatments. We suspect this technique will be successful in patients who have responded well to other therapies in all areas except for non-hair bearing areas.

DETAILED DESCRIPTION:
Vitiligo is an autoimmune skin condition that can have a profound psychosocial impact on patients. Vitiligo is caused by an immune-mediated destruction of melanocytes, or the cells responsible for producing melanin, which gives the skin its pigment. There are safe and effective treatments for vitiligo, which should be selected based on disease subtype, the percentage of body surface area involved, patient preference, and the impact of the disease on a patient's quality of life. Treatment aims to stabilize depigmented lesions, reduce disease progression and stimulate repigmentation. The current therapies available include topical and systemic immunosuppressants, phototherapy and surgical techniques.

The autologous transplantation of hair follicles has the ability to treat hairless areas by introducing follicular stem cells to an area of skin that would otherwise not respond to current treatment options. The potential to treat glabrous areas is of particular relevance for this technique, and the question proposed in this study is whether the same procedure of follicular hair transplant that has been previously safely and successfully used to treat segmental/stable vitiligo in hair bearing areas can applied to treat vitiligo in glabrous skin.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* Vitiligo patients already on treatment who demonstrate stable disease (have noted some repigmentation in hair bearing areas)
* Willingness to participate in the study
* Willingness to undergo biopsies of full-thickness skin tissue from areas without vitiligo and having them transplanted into areas with vitiligo
* Informed consent agreement signed by the subject

Exclusion Criteria:

* Adults unable to consent (adults lacking capacity)
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Unable to return for follow-up visits
* Infection or other dermatologic condition different than vitiligo in the area to be treated
* Personal or family history of keloid formation
* Known allergies to injectable lidocaine or other topical anesthetics
* Systemic immunosuppressive medication (oral corticosteroids) within prior 4 weeks
* Topical steroids at planned recipient site within the prior 1 week
* Individuals who are unwilling to discontinue topical steroids at recipient site
* Prescription or over-the-counter medication or cosmetics containing: retinoids, glycolic acid, salicylic acid, topical steroids at the site of treatment or oral corticosteroids, or any other remedies that might affect the healing process. Non-medicated moisturizers are allowed.
* Co-existent inflammatory skin disease
* Any other condition or laboratory value that would, in the professional opinion of the investigators, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with successful engraftment of hair follicles to transplant site | evaluated 10 days post-procedure visit
  Assessed by acceptance or rejection of graft into transplant site. Dermatologist will monitor for signs of rejection including infection, non-healing wounds, and necrosis of transplanted tissue and determine if transplant was successful (yes) or not (no), and the total percentage of successful cases will be calculated.
Percentage of repigmentation assessed by 4 point scale | evaluated at 3 month follow up visit
  Assessments of repigmentation will be performed by two dermatologists who will use photographs to determine percentage of repigmentation using the following scale: (excellent= 100%-95%, good= 94%-65%, fair= 64%-25%, poor= 24%-0%)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Rashighi, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No